CLINICAL TRIAL: NCT06852560
Title: GEM: A Single-Arm Trial Assessing Feasibility of Allostatic Load Biomarkers and CVD Risk Among Black Breast Cancer Survivors
Brief Title: A Trial Assessing Feasibility of Allostatic Load Biomarkers and CVD Risk Among Black Breast Cancer Survivors
Acronym: GEM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left institution
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UF-CCPS-0XX
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Black breast cancer survivors; allostatic load; atherosclerotic cardiovascular disease
MeSH Terms: conditions — Breast Neoplasms; Atherosclerosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gratitude, exercise and mindfulness program (Experimental)
  Interventions: Behavioral: Gratitude, exercise, and mindfulness program

INTERVENTIONS:
Behavioral: Gratitude, exercise, and mindfulness program — Participants will be enrolled in an 8-week GEM (Gratitude, Exercise, and Mindfulness) program conducted entirely in person at Blossoming Butterfly in Gainesville, Florida. Participants will attend weekly group sessions combining gratitude journaling, mindfulness-based stress reduction/emotional freedom technique, and physical activity goal-setting. Participants will also be provided with a toolkit to support at-home practices, including gratitude journaling, physical activity tracking, and mindfulness meditation.
  Blood, saliva and urine will be collected from each participant at baseline and post-intervention to measure the following allostatic load biomarkers: fasting glucose or hemoglobin A1c; lipid panel (total cholesterol, LDL, HDL); C-reactive protein; dehydroepiandrosterone sulfate; cortisol; glomerular filtration rate; and albumin-to-creatinine ratio.

SUMMARY:
This study's overall objective is to test the effects of a culturally tailored gratitude, exercise, and mindfulness/emotional freedom techniques (GEM) psychosocial intervention on allostatic load and atherosclerotic cardiovascular disease risk in black women breast Cancer survivors. Allostatic load refers to the cumulative physiological burden of chronic stress, which is a major contributor to CVD risk, impaired immune function, and worse cancer outcomes. Atherosclerotic cardiovascular disease risk encompasses factors such as blood pressure, cholesterol, and glucose control that predict long-term cardiovascular health.

Among survivors of breast cancer in the U.S., black women have the highest rates of mortality from breast cancer, cardiometabolic disease, and all causes. These disparities are likely due to complex interactions between socioeconomic, psychosocial, and biological risk factors. A higher prevalence of cardiometabolic risk factors among black women breast cancer survivors is one critical disparity associated with poorer breast cancer outcomes and increased cardiometabolic risk, including that driven by cardiotoxicity from breast cancer treatment. Engagement in physical activity, which reduces cardiometabolic risk, is associated with significant reductions in all-cause and cancer mortality in breast cancer survivors. However, black breast cancer survivors report lower levels of physical activity compared to their white counterparts, and most interventions targeting this behavior have not effectively engaged black women. Interventions that effectively increase physical activity in black women breast cancer survivors hold promise as a means for reducing these persistent disparities in survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must identify as Black women who have survived breast cancer
* Participants must have completed primary cancer treatment (surgery, chemotherapy, and/or radiation) at least 6 months prior to enrollment
* Adults ≥ 18 years old
* Capable of completing study requirements
* Informed consent obtained from the participant and documentation of participant agreement to comply with all study-related processes

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Impaired cognition (i.e., inability to follow and respond appropriately during screening).
* Participants currently enrolled in other lifestyle, exercise, or psychosocial interventions will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 8 months
  Determine the feasibility of collecting a comprehensive panel of allostatic load biomarkers and atherosclerotic cardiovascular disease risk components. This will be measured by the number of subjects who successfully complete the baseline assessments, which include self-reported questionnaires and biomarker collection, participate in a minimum number of 6 of 8 intervention sessions, and complete the post-intervention assessments, including follow-up questionnaires and biomarker collection.

SECONDARY OUTCOMES:
Difference in fasting glucose | 8 weeks
  Determine the difference in blood fasting glucose between baseline and post-intervention.
Difference in hemoglobin A1c | 8 weeks
  Determine the difference in blood hemoglobin A1c between baseline and post-intervention.
Difference in total cholesterol | 8 weeks
  Determine the difference in blood total cholesterol between baseline and post-intervention.
Difference in LDL | 8 weeks
  Determine the difference in blood LDL between baseline and post-intervention.
Difference in HDL | 8 weeks
  Determine the difference in blood HDL between baseline and post-intervention.
Difference in C-reactive protein | 8 weeks
  Determine the difference in blood C-reactive protein between baseline and post-intervention.
Difference in cortisol | 8 weeks
  Determine the difference in saliva cortisol between baseline and post-intervention.
Difference in glomerular filtration rate | 8 weeks
  Determine the difference in blood glomerular filtration rate between baseline and post-intervention.
Difference in albumin to creatinine ratio | 8 weeks
  Determine the difference in urine albumin to creatinine ratio between baseline and post-intervention.
Difference in Gratitude Questionnaire-6 score | 8 months
  Determine the difference in Gratitude Questionnaire-6 score between baseline and post-intervention.
Difference in International Physical Activity Questionnaire score | 8 months
  Determine the difference in International Physical Activity Questionnaire score between baseline and post-intervention.
Difference in The Gratitude Questionnaire-Six Item Form score | 8 months
  Determine the difference in The Gratitude Questionnaire-Six Item Form score between baseline and post-intervention.
Difference in Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACTIT-Sp) score | 8 months
  Determine the difference in FACTIT-Sp score between baseline and post-intervention.
Difference in General Self-Efficacy Scale score | 8 months
  Determine the difference in General Self-Efficacy Scale score between baseline and post-intervention.
Difference in Superwoman Schema score | 8 months
  Determine the difference in Superwoman Schema score between baseline and post-intervention.
Difference in Perceived Stress Scale score | 8 months
  Determine the difference in Perceived Stress Scale score between baseline and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lakeshia Cousin, PhD, APRN, Principal Investigator — University of Florida